CLINICAL TRIAL: NCT01277614
Title: A Randomized Control Trial for the Implementation of Lifestyle Modifications to Reduce the Burden of Chronic Disease Among University Staff
Brief Title: Therapeutic Lifestyle Modifications to Reduce Burden of Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Professor Dan Ramdath, The University of the West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMS-STA-08-01
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Metabolic Syndrome; Triglycerides; Blood Pressure; Diabetes
Keywords: lifestyle; diet; exercise
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): This is a 6-month intervention in which participants with 2 or more MS components are randomly assigned to intervention or control group. Intervention comprise individual diet counseling, an exercise plan and monthly lifestyle workshops. Controls receive printed material on healthy eating and lifestyle modification.
  Interventions: Behavioral: Therapeutic lifestyle
- Health Literature (Placebo Comparator)
  Interventions: Behavioral: Therapeutic lifestyle

INTERVENTIONS:
Behavioral: Therapeutic lifestyle — This is a 6-month intervention in which participants with 2r more MS components are randomly assigned to intervention or control group. Intervention comprise individual diet counseling, an exercise plan and monthly lifestyle workshops. Controls receive printed material on healthy eating and lifestyle modification.
  Other Names: diet counseling; exercise

SUMMARY:
The investigators previously established that there was a high burden of disease among all categories of staff at the University of the West Indies, St. Augustine and in many ways, this group is typical of the working class of the Caribbean population. Many had poor lifestyle behaviors, 23.8% had Metabolic Syndrome (MS) with many having one or more MS components. Since most time is spent at work, the workplace is understandably the most logical location to address issues pertaining to health, disease prevention and wellness and on-site programs have yielded many health and other benefits to employees and employers alike. Onwards of the 1980s, numerous studies have been done on work-site intervention programs and these have shown that if a company is able to identify employees at risk for developing health problems and then intervene, health risks and the resulting medical problems are reduced. Such a program, if tailored to meet the needs of participants, may yield similar benefits among the staff of the University of the West Indies.

DETAILED DESCRIPTION:
To conduct a randomized controlled intervention of lifestyle modifications among individuals with a high burden of metabolic syndrome components such as high body mass index, high fasting blood glucose and abnormal lipid profile.

A 6-month intervention is designed for implementation to detect a 20% reduction in MS components with 90% confidence. Participants (n=148) had 2 or more MS components and will be randomly assigned to intervention or control group. Intervention will comprise individual diet counseling, an exercise plan and monthly lifestyle workshops. Controls will receive printed material on healthy eating and lifestyle modification.

ELIGIBILITY:
Inclusion Criteria:

* having 2 or more metabolic syndrome components

Exclusion Criteria:

* having less than 2 metabolic syndrome components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
decrease waist circumference | 6 months
decrease fasting blood glucose | 6 months
decrease body mass index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Ramdath, PhD, Study Director — The University of The West Indies; Debbie G Hilaire, MSc, RD, Principal Investigator — The University of The West Indies
Locations (1):
- Dan Ramdath, Saint Augustine, Mount Hope, Trinidad and Tobago

REFERENCES:
- [Background] Ezenwaka CE, Nwagbara E, Seales D, Okali F, Sell H, Eckel J.Insulin resistance, leptin and monocyte chemotactic protein-1 levels in diabetic and non-diabetic Afro-Caribbean subjects.Arch Physiol Biochem. 2009 Feb;115(1):22-7. Ezenwaka CE, Nwagbara E, Seales D, Okali F, Hussaini S, Raja B, Wheeler V, Sell H, Avci H, Eckel J. A comparative study of the prevalence of the metabolic syndrome and its components in type 2 diabetic patients in two Caribbean islands using the new International Diabetes Federation definition. Arch Physiol Biochem. 2007 Oct-Dec;113(4-5):202-10. Ezenwaka CE.Serum lipid concentrations and Indices of obesity among adult subjects of the West Indies. Ann Saudi Med. 2002 Jan-Mar;22(1-2):112-4. Ezenwaka CE, Offiah NV.Differences in cardiovascular disease risk factors in elderly and younger patients with type 2 diabetes in the West Indies. Singapore Med J. 2002 Oct;43(10):497-503. Ezenwaka CE, Kalloo R.Indices of obesity, dyslipidemia, and insulin resistance in apparently healthy Caribbean subjects. J Clin Lab Anal. 2003;17(1):6-11.